CLINICAL TRIAL: NCT03834688
Title: Phase II Study of Bendamustine and Rituximab Plus Venetoclax in Untreated Mantle Cell Lymphoma Over 60 Years of Age
Acronym: PrE0405
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PrE0405; ML40551 (Other: Genentech)
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: Venetoclax; Bendamustine; Rituximab; Bcl-2 Family Protein Inhibitor
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — venetoclax; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Intervention Model Description: Open-Label, Single-Arm Study, Cycle 1 Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction (Experimental): Venetoclax, bendamustine and rituximab as induction therapy for 6 cycles of 28 days.
  Interventions: Drug: Venetoclax; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Venetoclax — Cycle 1: Venetoclax by mouth daily. The dose will gradually increase during Cycle 1. (Day 1-7: 20 mg; Day 8-14: 50 mg; Day 15-21: 100 mg; Day 22-28: 200 mg.)
  Cycles 2-6: Venetoclax 400 mg by mouth daily on Days 1-10 (1 cycle = 28 days).
  Other Names: GDC-0199; ABT-199; RO5537382
Drug: Bendamustine — Cycle 1-6: Bendamustine 90 mg/m² intravenous (IV) on Days 1 and 2 of each cycle. Bendamustine may be started at 70 mg/m² in patients over the age of 75 years with comorbid conditions or patients over the age of 80 years without comorbid conditions.
  Other Names: Bendamustine hydrochloride
Drug: Rituximab — Cycle 1-6: Rituximab 375 mg/m² IV on Day 1 of each cycle. After 2 consecutive cycles of Rituximab IV are well tolerated, Rituximab may be given subcutaneously.
  Other Names: Chimeric anti-CD20 monoclonal antibody; Rituxan

SUMMARY:
Eligible untreated patients will receive single arm venetoclax, bendamustine and rituximab as induction therapy. After 6 cycles, maintenance rituximab may be administered per physician discretion.

Venetoclax is an oral Bcl-2 family protein inhibitor. It targets the B-cell lymphoma 2 (BCL-2) protein, which supports cancer cell growth and is overexpressed in many patients with mantle cell lymphoma. Venetoclax may make the cancer cells sensitive to chemotherapy. This may help to slow down the growth of cancer or may cause cancer cells to die.

The purpose of this study is to see if venetoclax in combination with bendamustine and rituximab chemotherapy is effective in treating people who have mantle cell lymphoma and to examine the side effects, good and bad, associated with this combination.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is a subtype of Non-Hodgkin Lymphoma (NHL) which is considered incurable with conventional therapy. With an incidence of approximately 70,000 cases diagnosed in the United States (US) per year, the disease is rare.

This is an open-label phase II study of venetoclax in combination with bendamustine and rituximab. Patients will receive induction therapy with venetoclax, bendamustine and rituximab for six cycles (1 cycle = 28 days). There will be an interim analysis after 19 patients are enrolled to evaluate for tumor lysis syndrome (TLS). TLS is caused by the fast breakdown of cancer cells which can lead to electrolyte and kidney problems.

Tumor assessments will be performed after Cycle 3-4 and at end of induction therapy.

Mandatory pre-treatment tumor tissue sample (i.e., obtained in the course of standard biopsy or surgery) will be required for research (if sufficient tissue is available).

Mandatory bone marrow aspirate (obtained in the course of standard biopsy) and peripheral blood sample will be collected at the end of treatment for Minimal Residual Disease (MRD). MRD measures the disease remaining after treatment. Optional peripheral blood samples will also be collected for future research.

10/11/2021: Due to slower than anticipated enrollment, the study was redesigned to reflect the current historical complete response rate and with a lowered sample size for prompt primary endpoint readout.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed (biopsy-proven) diagnosis of mantle cell lymphoma (MCL), with documented cyclin D1 (BCL1) expression by immunohistochemical stains and/or t(11;14) by cytogenetics or Fluorescence In Situ Hybridization (FISH).
* Patients must have measurable or evaluable disease as defined as a lymph node measuring >1.5 cm in any dimension or splenomegaly with spleen >15 cm in craniocaudal dimension.
* Age ≥ 60 years.
* No intention to undergo consolidation with high dose chemotherapy and autologous stem cell rescue (Autologous Stem Cell Transplant) in first remission.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Ability to understand and willingness to sign Institutional Review Board (IRB)-approved informed consent.
* Willing to provide mandatory tissue samples (if sufficient tissue available), bone marrow and blood samples for research purposes.
* Adequate organ function as measured by the following criteria, obtained ≤ 2 weeks prior to registration:

  * Absolute Neutrophil Count (ANC) ≥ 1000/mm³
  * Hemoglobin ≥ 8 g/dL
  * Platelets ˃75,000/mm³
  * Creatinine clearance ≥ 40 mL/min, calculated with the use of 24-hour creatinine clearance or by Cockcroft-Gault formula
  * Total Bilirubin ≤ 1.5x Upper Limit of Normal (ULN) or ≤ 3x ULN for patients with documented Gilbert's syndrome
  * Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 2.5x ULN
* All females of childbearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have a blood test to rule out pregnancy within 2 weeks prior to registration.
* Women must not be pregnant or breastfeeding. Females of childbearing potential who are sexually active with a non-sterilized male partner and sexually active men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) prior to study entry, for the duration of study participation, and for 12 months after last dose of therapy. Method of contraception must be documented.
* Patients should not have prior chemotherapy, radiotherapy or immunotherapy for lymphoma.
* Patients must have no recent (<1 year) history of malignancy except for the following:

  * adequately treated non-melanoma skin cancer
  * adequately treated Stage I melanoma of the skin
  * in situ cervical cancer
  * low grade prostate adenocarcinoma (Gleason grade ≤ 6) managed with observation and stable for 6 months.
* Patients should not have known evidence of central nervous system (CNS) lymphoma.
* Patients must not have received a prior allogeneic stem cell transplant or solid organ transplant (except for cornea) for any indication.
* Patients must have no active, uncontrolled infections.
* Patients must not have active hepatitis B or be chronic carriers of hepatitis B. This is defined as patients with hepatitis B surface antigen (HBsAg) positive. Patients with prior exposure to hepatitis B (hepatitis B core antibody (anti-HBc) positive AND HBsAg negative) are allowed with a protective level hepatitis B surface antibody AND a negative hepatitis B viral load by polymerase-chain reaction (PCR).
* Patients must not have active hepatitis C (HCV) as defined by a hepatitis C viral load detectable by PCR. Patients with a negative HCV antibody are assumed to have a negative HCV viral load. Patients with a positive HCV antibody must have a negative hepatitis C viral load by PCR. Prior treatment for an active HCV infection will be allowed as long as the hepatitis C viral load by PCR is negative.
* Patients must not have known active Human Immunodeficiency Virus (HIV). Testing not required in absence of clinical suspicion.
* Patients must not have evidence of significant, uncontrolled concomitant diseases, including psychiatric diseases, that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient.
* Patients must not have conditions that preclude oral administration or absorption of medications through the GI tract, including but not limited to the inability to swallow pills or malabsorption syndromes.
* Patients must not have known allergies to both xanthine oxidase inhibitors and rasburicase.
* Patients must not require the use of warfarin. Blood thinners of other classes are permitted.
* Patient may not receive the following agents within 7 days prior to the first dose of venetoclax:

  * Strong and moderate CYP3A inhibitors
  * Strong and moderate CYP3A inducers
  * Strong and moderate P-gp inhibitors
* Patients must not have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Portell, MD, Study Chair — University of Virginia
Locations (7):
- United States (7):
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - St. Joseph Mercy Hospital Cancer Care Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
Data is proprietary

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction: Venetoclax, bendamustine and rituximab as induction therapy for 6 cycles of 28 days.
  Venetoclax: Cycle 1: Venetoclax by mouth daily. The dose will gradually increase during Cycle 1. (Day 1-7: 20 mg; Day 8-14: 50 mg; Day 15-21: 100 mg; Day 22-28: 200 mg.)
  Cycles 2-6: Venetoclax 400 mg by mouth daily on Days 1-10 (1 cycle = 28 days).
  Bendamustine: Cycle 1-6: Bendamustine 90 mg/m² intravenous (IV) on Days 1 and 2 of each cycle. Bendamustine may be started at 70 mg/m² in patients over the age of 75 years with comorbid conditions or patients over the age of 80 years without comorbid conditions.
  Rituximab: Cycle 1-6: Rituximab 375 mg/m² IV on Day 1 of each cycle. After 2 consecutive cycles of Rituximab IV are well tolerated, Rituximab may be given subcutaneously.
Period: Overall Study
Arm/Group | Induction
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 30
Age, Continuous [Median (Full Range); unit: years] | 71 [61 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). A score of 0 indicates fully active, 1 indicates restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2 indicates ambulatory and capable of all selfcare but unable to carry out any work activities, 3 indicates capable of only limited selfcare, and 4 indicates completely disabled.
  Participants
    0 | 9
    1 | 21
    2 | 3
Mantle Cell Lymphoma (MCL) International Prognostic Index (MIPI) Risk Category [Count of Participants; unit: Participants] — Mantle Cell Lymphoma (MCL) International Prognostic Index (MIPI) is a commonly used risk stratification score that classifies patients with MCL into low-, intermediate-, and high-risk groups for overall survival. Prognosis is worst in the high-risk category.
  Participants
    Low risk | 2
    Intermediate risk | 9
    High risk | 22

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate at End of Induction
Description: Complete Response (CR) was assessed in accordance with the Lugano Classification Criteria using PET/CT scans (at baseline) and PET/CT or CT scans (during follow-up). Based on this criteria, a Deauville score ≤ 3 corresponds to a CR, a score of 4 or 5 and ≥ 50% decrease in the sum of lesion measurements corresponds to a Partial Response (PR), a score of 4 or 5 and <50% decrease in sum of lesion measurements corresponds to a Stable Disease (SD), a score of 4 or 5 and >1.5cm increase in a single lesion or presence of new lesions or bone marrow recurrence denotes Progressive Disease (PD).
Time Frame: Complete Response (CR) status was assessed after 6 months of induction treatment, plus an additional 2 months for end of treatment PET/CT scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction
Number analyzed (Participants) | 33
Participants
  Complete response | 28
  Partial response | 4
  Stable disease | 0
  Progressive disease | 0
  Unevaluable | 1

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Number of participants with abnormal laboratory values and/or adverse events including Tumor Lysis Syndrome (TLS) were assessed using CTCAE v5.0. The adverse events were graded on a scale of 1 to 5 based on severity: grade 1 is mild, grade 2 is moderate, grade 3 is severe, grade 4 is life-threatening, and grade 5 resulted in death.
Time Frame: Adverse events were reported throughout 6 months of induction treatment and up to 2 months following completion of induction treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Induction
Number analyzed (Participants) | 33
Participants
  Grade 1 | 5
  Grade 2 | 8
  Grade 3 | 11
  Grade 4 | 6
  Grade 5 | 2
  No treatment-related AE | 1

3. Secondary Outcome: Overall Response
Description: Objective response was assessed in accordance with the Lugano Classification Criteria using PET/CT scans (at baseline) and PET/CT or CT scans (during follow-up). Objective response is defined as the number of patients with a best treatment response of complete (CR) or partial response (PR).
Time Frame: Objective response was assessed after 6 months of induction treatment, plus an additional 2 months for end of treatment PET/CT scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction
Number analyzed (Participants) | 33
Participants
  Complete or partial response | 32
  Stable or progressive disease, or unevaluable | 1

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is a measure of patients that are alive and progression-free. Survival status is ascertained via direct contact and disease progression was assessed in accordance with the Lugano Classification Criteria using PET/CT scans (at baseline) and PET/CT or CT scans (during follow-up).
Time Frame: Progression-Free Survival (PFS) was assessed from the start to completion of induction treatment (6 months) through the completion of maintenance treatment (24 months) for up to 48 months. PFS at the 4-year timepoint was estimated and reported.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction
Number analyzed (Participants) | 33
Percentage of Participants | 59.0 [33.7 to 77.5]

5. Secondary Outcome: Overall Survival (OS)
Description: Patients' survival status was measured by direct contact. The proportion of patients that are alive at the 4-year study timepoint is reported.
Time Frame: Overall survival (OS) was assessed from the start to completion of induction treatment (6 months) through the completion of maintenance treatment (24 months) for up to 48 months. OS at the 4-year timepoint was estimated and reported.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction
Number analyzed (Participants) | 33
Percentage of Participants | 61.3 [36.2 to 79.0]

ADVERSE EVENTS:
Time Frame: Patients were followed for up to 48 months, which covers 6 months of induction treatment and 24 months of maintenance treatment.
Arm/Group | Induction
All-Cause Mortality (participants affected / at risk) | 10/33
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 19/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (N=33)
COVID-19 pneumonia (Infections and infestations) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (N=33)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 9 (12)
Neutropenia (Investigations) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
White blood cell count decreased (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03834688/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03834688/SAP_001.pdf